CLINICAL TRIAL: NCT00886821
Title: A Phase 1, Placebo-controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Escalating Subcutaneous Doses Of Cvx-096 In Type 2 Diabetic Adult Subjects
Brief Title: A Safety and Pharmacokinetic Study of CVX-096 in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1111001; CVX-096-101 (Other: Alias Study Number)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 1 Type 2 diabetes CVX-096 diabetes mellitus; adult-onset diabetes mellitus; non-insulin dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: CVX-096

INTERVENTIONS:
Biological: CVX-096 — Subcutaneous administration of CVX-096 with doses ranging from 0.1 mg up to a maximum of 36 mg

SUMMARY:
The purpose of this study is to determine safety and tolerability of CVX-096 in adult, type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients (females will be women of non-childbearing potential) with an historical diagnosis of type 2 diabetes mellitus, who are currently being treated with metformin at a dose at or near maximum.
* Hb A1c between 7-10%.
* Fasting C-peptide >0.4 nmol/L.

Exclusion Criteria:

* History of clinically significant chronic conditions other than T2DM not well controlled by either diet or medications.
* Patients with pancreatitis or considered a high risk for pancreatitis.
* History of contraindications to metformin therapy.
* Previous treatment with an approved or investigational GLP 1 mimetic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Cetero Research, Miami Gardens, Florida
  - Cetero Research - San Antonio, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1111001&StudyName=A%20Safety%20and%20Pharmacokinetic%20Study%20of%20CVX-096%20in%20Type%202%20Diabetics%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consist of two stages: stage 1 and stage 2. Participants were enrolled and randomized for stage 1 and stage 2 separately.
Groups:
- Cohort 1: PF-04856883 0.1 Milligram (mg): Participants received single subcutaneous injection of PF-04856883 (CVX-096) 0.1 mg on Day 1.
- Cohort 2: PF-04856883 0.3 mg: Participants received single subcutaneous injection of PF-04856883 0.3 mg on Day 1.
- Cohort 3: PF-04856883 1.0 mg: Participants received single subcutaneous injection of PF-04856883 1.0 mg on Day 1.
- Cohort 4: PF-04856883 3.0 mg: Participants received single subcutaneous injection of PF-04856883 3.0 mg on Day 1.
- Cohort 5: PF-04856883 6.0 mg: Participants received single subcutaneous injection of PF-04856883 6.0 mg on Day 1.
- Cohort 6: PF-04856883 12.0 mg: Participants received single subcutaneous injection of PF-04856883 12.0 mg on Day 1.
- Cohort 7: PF-04856883 24.0 mg: Participants received single subcutaneous injection of PF-04856883 24.0 mg on Day 1.
- Cohort 8: PF-04856883 36.0 mg: Participants received single subcutaneous injection of PF-04856883 36.0 mg on Day 1.
- Cohort 9: PF-04856883 18.0 mg: Participants received subcutaneous injection of PF-04856883 18.0 mg on Day 1 and 8.
- Cohort 1-9: Placebo: Participants received placebo matched to PF-04856883 subcutaneous injection either single dose on Day 1 or multiple dose on Day 1 and 8 respectively.
- Cohort 10: PF-04856883 15.0 mg: Participants received subcutaneous injection of PF-04856883 15.0 mg on Day 1, 8, 15 and 22.
- Cohort 11: PF-04856883 20.0 mg: Participants received subcutaneous injection of PF-04856883 20.0 mg on Day 1, 8, 15 and 22.
- Cohort 12: PF-04856883 25.0 mg: Participants received subcutaneous injection of PF-04856883 25.0 mg on Day 1, 8, 15 and 22.
- Cohort 10-12: Placebo: Participants received placebo matched to PF-04856883 subcutaneous injection on Day 1, 8, 15 and 22.
Period: Stage 1
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Started | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 18 | 0 | 0 | 0 | 0
Completed | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 18 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 13 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Groups:
- Cohort 9: Placebo: Participants received placebo matched to PF-04856883 subcutaneous injection either single dose on Day 1 or two dose on Day 1 and 8 respectively.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 18 | 9 | 9 | 13 | 9 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 6 | 7 | 6 | 5 | 5 | 4 | 5 | 13 | 8 | 8 | 13 | 8 | 101
  >=65 years | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5 | 1 | 1 | 0 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 5 | 3 | 2 | 5 | 6 | 0 | 3 | 4 | 4 | 3 | 0 | 39
  Male | 7 | 3 | 5 | 2 | 3 | 4 | 1 | 0 | 6 | 15 | 5 | 5 | 10 | 9 | 75

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-04856883 on Day 1
Description: AUClast was defined as area under the concentration-time curve from time zero to the time of last measured concentration and calculated by using linear up/log down trapezoidal method.
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose on Day 1
Population: Pharmacokinetic (PK) analysis population included all randomized participants who received at least 1 dose of PF-04856883 and had PK data. 'N'(Overall number of participants)=participants who were evaluable for this outcome measure. This outcome measure was not planned to be analyzed in multiple dosing cohort(Cohort 9),as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr)/mL
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr)/mL | 865 (625.3) | 4960 (462.0) | 7065 (192.1) | 32552 (127.7) | 105950 (53.4) | 304167 (25.9) | 120521 (5404.6) | 297503 (211.1)

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04856883 on Day 1
Time Frame: Cohort 1-9: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose on Day 1; Cohort 10-12: pre-dose, 1 and 6 hours post-dose on Day 1
Population: PK analysis population included all randomized participants who received at least 1 dose of PF-04856883 and had PK data. Here, 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 13
hour | 156 [144 to 168] | 72.1 [36.0 to 144] | 168 [96.0 to 168] | 72.0 [48.0 to 168] | 144 [72.0 to 168] | 120 [72.0 to 168] | 108 [36.0 to 168] | 96.0 [48.0 to 168] | 84.0 [36.0 to 144] | 168 [48.0 to 168] | 168 [48.0 to 168] | 168 [25.1 to 194]

3. Primary Outcome: Stage 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04856883 on Day 8
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose on Day 8
Population: PK analysis population included all randomized participants who received at least 1 dose of PF-04856883 and had PK data. The outcome was not planned to be analyzed for single dosing cohorts (Cohort 1 to 8), since the dosing was done only on Day 1 in these cohorts.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 9: PF-04856883 18.0 mg
Number analyzed (Participants) | 6
hour | 72.0 [48.0 to 96.0]

4. Primary Outcome: Stage 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04856883 on Day 22
Time Frame: pre-dose, 1 and 6 hours post-dose on Day 22
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg
Number analyzed (Participants) | 9 | 7 | 7
hour | 48.0 [6.00 to 168] | 46.9 [1.00 to 48.0] | 48.0 [47.2 to 168]

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04856883 on Day 1
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 13
nanogram per milliliter (ng/mL) | 7.05 (104.9) | 29.0 (126.3) | 24.8 (92.3) | 149 (63.2) | 387 (52.4) | 900 (36.2) | 579 (1314.6) | 1299 (104.3) | 1082 (50.0) | 736 (47.1) | 1554 (38.3) | 958 (63.1)

6. Primary Outcome: Stage 1: Maximum Observed Plasma Concentration (Cmax) of PF-04856883 on Day 8
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose on Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 9: PF-04856883 18.0 mg
Number analyzed (Participants) | 6
ng/mL | 1536 (54.9)

7. Primary Outcome: Stage 2: Maximum Observed Plasma Concentration (Cmax) of PF-04856883 on Day 22
Time Frame: pre-dose, 1 and 6 hours post-dose on Day 22
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg
Number analyzed (Participants) | 9 | 8 | 7
ng/mL | 1767 (37.6) | 2193 (36.9) | 2253 (31.9)

8. Secondary Outcome: Stage 1: Apparent Terminal Elimination Half-Life (t1/2) of PF-04856883 on Day 1
Description: Apparent terminal elimination half-life is the time measured for the plasma concentration of PF-04856883 to decrease by one-half of its initial concentration.
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose on Day 1
Population: PK analysis population included all randomized participants who received at least 1 dose of PF-04856883 and had PK data. Here, 'N' signifies those participants who were evaluable for this outcome measure. This outcome measure was not planned to be analyzed in multiple dosing cohort (Cohort 9), as pre specified in protocol.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 5 | 6 | 5 | 4
hour | NA (NA) — Data was not estimable since PK concentration was below the lower limit of quantification. | 188 (42.6) | 151 (5.14) | 186 (53.3) | 144 (12.0) | 163 (52.0) | 156 (45.6) | 159 (37.5)

9. Secondary Outcome: Stage 1: Apparent Terminal Half-Life (t1/2) of PF-04856883 on Day 8
Description: as for outcome 8
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 9: PF-04856883 18.0 mg
Number analyzed (Participants) | 6
hour | 156 (23.4)

10. Secondary Outcome: Stage 2: Apparent Terminal Elimination Half-Life (t1/2) of PF-04856883 on Day 22
Description: as for outcome 8
Time Frame: pre-dose, 1 and 6 hours post-dose on Day 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg
Number analyzed (Participants) | 8 | 8 | 5
hour | 156 (32.7) | 102 (44.9) | 149 (29.0)

11. Secondary Outcome: Stage 1: Mean Residence Time (MRT) of PF-04856883 on Day 1
Description: MRT is defined as AUMC(0 - inf) divided by AUC(0 - inf), where AUMC(0 - inf) is the area under the first moment curve from time 0 extrapolated to infinite time, calculated using the linear/log trapezoidal method and AUC(0 - inf) is the area under the concentration-time curve extrapolated to infinity.
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose Day 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 5 | 6 | 5 | 4
hour | NA [NA to NA] — Data was not estimable since PK concentration was below the lower limit of quantification. | 310 (69.4) [205 to 373] | 316 (20.3) [286 to 325] | 350 (70.5) [227 to 399] | 281 (31.6) [217 to 295] | 319 (77.8) [176 to 390] | 239 (89.7) [189 to 414] | 312 (70.7) [216 to 378]

12. Secondary Outcome: Stage 1: Apparent Oral Clearance (CL/F) of PF-04856883 on Day 1
Description: Apparent oral clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug apparent oral clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose Day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 5 | 6 | 5 | 4
Liter per hour (L/hr) | NA (NA) — Data was not estimable since PK concentration was below the lower limit of quantification. | 0.0176 (20.4) | 0.0643 (27.4) | 0.0562 (36.5) | 0.0487 (53.5) | 0.0354 (25.6) | 0.0530 (47.5) | 0.0527 (28.6)

13. Secondary Outcome: Stage 1: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC[0 - Inf]) of PF-04856883 on Day 1
Description: AUC(0 - inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It was calculated as AUC (0-t) plus (last measurable concentration divided by apparent terminal elimination rate constant).
Time Frame: pre-dose, 1, 6, 18, 24, 36, 48, 72, 96, 144, and 168 hours post-dose Day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 5 | 6 | 5 | 4
L/hr | NA (NA) — Data was not estimable since PK concentration was below the lower limit of quantification. | 17013 (20.4) | 15550 (27.4) | 53420 (36.5) | 123081 (53.5) | 339062 (25.6) | 452842 (47.5) | 682543 (28.6)

14. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Cohort 1-8: Baseline up to Day 29; Cohort 9: Baseline up to Day 36; Cohort 10-12: Baseline up to Day 50
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 18 | 9 | 9 | 13 | 9
Participants
  AEs | 2 | 2 | 5 | 1 | 2 | 4 | 5 | 6 | 3 | 4 | 5 | 7 | 8 | 4
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Stage 1: Change From Baseline in Post-Prandial Area Under the Curve (AUC) of Glucose at Day 3 and 7
Description: Area under the glucose concentration-time curve from 0 minute (approximately 20 minutes prior to the meal) to 180 minutes post initiation of meal.
Time Frame: Baseline, Day 3 and 7
Population: Pharmacodynamic analysis population included all randomized participants who had received at least 1 dose of study medication and had PD data. Here, number analyzed signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: milligram*hour per deciliter (mg*hr)/dL
Groups:
- Cohort 1-8: Combined Placebo: Participants received placebo matched to PF-04856883 subcutaneous injection on Day 1, 3, 7.
- Cohort 9: Placebo: Participants received placebo matched to PF-04856883 subcutaneous injection either single dose on Day 1 or multiple dose on Day 1 and 8 respectively.
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2
milligram*hour per deciliter (mg*hr)/dL
  Change at Day 3: number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 0 | 15 | 0
  Change at Day 3 | 1.44 (102) | 44.9 (76.8) | -92.3 (78.2) | -54.0 (60.0) | 46.7 (70.9) | -74.5 (59.7) | -140 (124) | -80.1 (70.6) |  | -10.6 (95.3) |
  Change at Day 7 | -38.8 (95.5) | 29.3 (161) | -147 (93.4) | -23.0 (125) | 65.1 (85.1) | -39.6 (52.6) | -108 (139) | -38.4 (66.7) | -119 (81.7) | -9.04 (119) | -46.1 (6.98)

16. Other Pre Specified Outcome: Stage 1: Change From Baseline in 7-point Weighted Mean Glucose at Day 3 and Day 7
Description: It was assessed by 7-point glucose measurements via the glucose oxidase method.
Time Frame: Baseline, Day 3 and 7
Population: Pharmacodynamic analysis population included all randomized participants who had received at least 1 dose of study medication and had PD data.
Measure: Mean (Standard Deviation); unit: milligram per deciliter(mg/dL)
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2
milligram per deciliter(mg/dL)
  Change at Day 3 | 3.27 (24.1) | -0.0252 (16.3) | -17.9 (21.7) | 1.04 (18.2) | 20.2 (18.4) | -15.7 (12.4) | -31.7 (30.5) | -26.4 (22.9) | -23.9 (10.6) | 0.506 (25.0) | -16.6 (12.0)
  Change at Day 7 | -15.6 (23.0) | 7.44 (42.1) | -28.7 (26.9) | -8.45 (33.6) | 7.05 (53.2) | -20.5 (10.2) | -33.9 (42.1) | -24.4 (29.4) | -12.8 (29.8) | -5.22 (25.9) | -23.0 (11.0)

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Hemoglobin (Hgb), hematocrit: less than (<) 0.8*lower limit of normal (LLN), platelet: <75 or greater than (>) 700*10^3/millimeter (mm)^3*upper limit of normal (ULN), leukocyte: <2.5 or >17.5*10^3/mm^3*ULN; total bilirubin 1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase: >3.0*ULN, total protein, albumin: <0.8*LLN or >1.2*ULN ;blood urea nitrogen, creatinine: >1.3*ULN, uric acid >1.2*ULN; sodium <0.95*LLN or >1.05*ULN, potassium, calcium: <0.9*LLN or >1.1*ULN, albumin, total protein <0.8*LLN or >1.2*ULN; glucose <0.6*LLN or >1.5*ULN, creatine kinase >2.0*ULN; urine (red blood cell, white blood cell >6/high power field).
Time Frame: Cohort 1-8: Baseline up to Day 28; Cohort 9: Baseline up to Day 35; Cohort 10-12; Baseline up to Day 50
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2 | 9 | 9 | 13 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Criteria for vital signs: pulse rate <40 beats per minute (bpm), supine, sitting and erect pulse rate <40 bpm, supine pulse rate >120 bpm, sitting pulse rate >120 bpm, and erect pulse rate >120 bpm; systolic blood pressure: SBP <90 millimeters of mercury (mmHg), change from baseline in SBP greater than or equal to (>=) 30 mmHg; diastolic blood pressure: DBP <50 mmHg, change from baseline in DBP >=20 mmHg.
Time Frame: Cohort 1-8: Baseline up to Day 28; Cohort 9: Baseline up to Day 35; Cohort 10-12; Baseline up to Day 50
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2 | 9 | 9 | 13 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Other Pre Specified Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Criteria for ECG findings: PR interval >=300 millisecond (msec), >=25 percent increase when baseline >200 msec, and >=50 percent increase when baseline less than or equal to (<=) 200 msec; QRS interval >=200 msec, >=25 percent increase when baseline >=100 msec, and >=50 percent increase when baseline <=100 msec; QT/QTc interval (corrected QT interval) >=500 msec.
Time Frame: Cohort 1-8: Baseline up to Day 28; Cohort 9: Baseline up to Day 35; Cohort 10-12; Baseline up to Day 50
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2 | 9 | 9 | 13 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: Number of Participants With Clinically Significant Physical Examinations
Description: Full physical examination included examination of the skin, eyes, ears, throat, neck, and cardiac, respiratory, gastrointestinal and musculoskeletal systems. The examination assessed the participants for any clinically significant changes in physical status, as determined by the investigator.
Time Frame: Cohort 1-8: Baseline up to Day 28; Cohort 9: Baseline up to Day 35; Cohort 10-12; Baseline up to Day 50
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2 | 9 | 9 | 13 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Other Pre Specified Outcome: Stage 1: Number of Participants With Hypoglycemia
Description: Blood glucose level was checked for hypoglycemia by glucometer. Criteria for hypoglycemia: blood glucose level <60 mg/dL if accompanied by symptoms, blood glucose level <=50 mg/dL regardless of symptoms.
Time Frame: Day 1: 0 hour (pre-dose) up to 48 hours post dose
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Other Pre Specified Outcome: Stage 1: Number of Participants With Clinically Significant Abnormal Rhythms
Description: Criteria for abnormal rhythms: asymptomatic marked sinus bradycardia rate <35 bpm; asymptomatic supraventricular couplets, atrial bigeminy lasting >30 seconds; asymptomatic ventricular couplets, ventricular bigeminy lasting >30 seconds; asymptomatic type I second degree (wenckebach) atrioventricular block of >30 seconds duration; asymptomatic frequent premature ventricular complexes (=>200/24 hours); asymptomatic frequent premature atrial complexes (=>240/24 hours).
Time Frame: Cohort 1- 8: Day 1 up to Day 3; Cohort 9: Day 1 up to Day 10
Population: Safety population will consist of all randomized patients who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Other Pre Specified Outcome: Stage 1: Number of Participants With Anti-Drug Antibodies
Time Frame: Day 0, 8, 14, 15, 21, 28 and 35
Population: Safety population included all randomized participants who received at least 1 dose of study medication. Here, number analyzed signifies those participants who were evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-8: Combined Placebo | Cohort 9: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 16 | 2
Participants
  Day 0 | 1 | 2 | 1 | 3 | 1 | 1 | 3 | 2 | 1 | 1 | 0
  Day 8 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 2 | 0 | 1 | 0
  Day 14: number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 0 | 16 | 0
  Day 14 | 0 | 2 | 2 | 2 | 1 | 1 | 3 | 2 |  | 1 |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2
  Day 15 |  |  |  |  |  |  |  |  | 0 |  | 0
  Day 21 | 0 | 2 | 1 | 2 | 1 | 2 | 4 | 2 | 1 | 1 | 0
  Day 28: number analyzed (Participants) | 7 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 0 | 16 | 0
  Day 28 | 0 | 2 | 1 | 2 | 1 | 1 | 4 | 2 |  | 1 |
  Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2
  Day 35 |  |  |  |  |  |  |  |  | 0 |  | 0

24. Other Pre Specified Outcome: Stage 2: Number of Participants With Anti-Drug Antibodies
Time Frame: Day 0, 29 and 50
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Number analyzed (Participants) | 9 | 9 | 13 | 9
Participants
  Day 0 (n= 9, 9, 13 ,9) | 1 | 1 | 2 | 0
  Day 29 (n= 9, 8, 7, 8): number analyzed (Participants) | 9 | 8 | 7 | 8
  Day 29 (n= 9, 8, 7, 8) | 0 | 1 | 2 | 0
  Day 50 (n= 9, 8, 8, 8): number analyzed (Participants) | 9 | 8 | 8 | 8
  Day 50 (n= 9, 8, 8, 8) | 0 | 3 | 3 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1: PF-04856883 0.1 Milligram (mg) | Cohort 2: PF-04856883 0.3 mg | Cohort 3: PF-04856883 1.0 mg | Cohort 4: PF-04856883 3.0 mg | Cohort 5: PF-04856883 6.0 mg | Cohort 6: PF-04856883 12.0 mg | Cohort 7: PF-04856883 24.0 mg | Cohort 8: PF-04856883 36.0 mg | Cohort 9: PF-04856883 18.0 mg | Cohort 1-9: Placebo | Cohort 10: PF-04856883 15.0 mg | Cohort 11: PF-04856883 20.0 mg | Cohort 12: PF-04856883 25.0 mg | Cohort 10-12: Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/18 | 0/9 | 0/9 | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 2/7 | 2/6 | 5/6 | 1/7 | 2/6 | 4/6 | 5/6 | 6/6 | 3/6 | 4/18 | 5/9 | 7/9 | 8/13 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-04856883 0.1 Milligram (mg) (N=7) | Cohort 2: PF-04856883 0.3 mg (N=6) | Cohort 3: PF-04856883 1.0 mg (N=6) | Cohort 4: PF-04856883 3.0 mg (N=7) | Cohort 5: PF-04856883 6.0 mg (N=6) | Cohort 6: PF-04856883 12.0 mg (N=6) | Cohort 7: PF-04856883 24.0 mg (N=6) | Cohort 8: PF-04856883 36.0 mg (N=6) | Cohort 9: PF-04856883 18.0 mg (N=6) | Cohort 1-9: Placebo (N=18) | Cohort 10: PF-04856883 15.0 mg (N=9) | Cohort 11: PF-04856883 20.0 mg (N=9) | Cohort 12: PF-04856883 25.0 mg (N=13) | Cohort 10-12: Placebo (N=9)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 5 | 1 | 0 | 2 | 2 | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 1 | 5 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 6 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.